CLINICAL TRIAL: NCT06439030
Title: Examining the Impact of a Mobile and Web-Based Healing Program on University Students Affected by Earthquakes and Experiencing High Levels of Trauma
Brief Title: Mobile and Web-Based Healing Program on University Students Affected by Earthquakes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Pınar Soylar, Associate Professor, Head of Nursing Department, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FiratU-PSOYLAR-001
Record Dates: First submitted 2024-05-03; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Trauma; Stress
Keywords: earthquake; Post-traumatic stress; Psychosocial support
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery group (Experimental): This is the group to which the interventions in the recovery program are applied.
  Interventions: Behavioral: Recovery program
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Recovery program — The practices included in the program are: Cinema Film Screening and Emotion/Thought Sharing, Laughter Yoga Practice, Stress Coping Techniques Training, Progressive Relaxation, Loss/Mourning Process Training, Expressive Art Therapy Practice, Healthy Lifestyle Behaviors Training.
  Arms: Recovery group

SUMMARY:
This research is a randomized controlled study that will be conducted in an online environment. The study comprises five stages. The first stage, PREPARATION, involves obtaining ethical approval and permissions from universities, preparing data collection tools, and identifying scholarship recipients. The second stage is the development of the MOBILE AND WEB-BASED application. The third stage is the SITUATION ASSESSMENT stage. In this stage, the post-earthquake trauma level, coping skill level, emotional eating levels, and the status of healthy lifestyle behavior of students enrolled in the Nursing Departments of firat University, Osmaniye Korkut Ata University, and Ankara University will be determined using one of the quantitative data collection tools, PETLDS (Objectives 1, 2, 3, and 4). The fourth stage is the INTERVENTION stage, where the prepared training and applications will be implemented within the program (Objectives 5, 6, 7, and 8). The fifth stage is the EVALUATION stage, involving the collection of final test data and analysis.

DETAILED DESCRIPTION:
The aim of this research is to investigate the effect of a mobile and web-based recovery program applied to university students affected by post-disaster earthquakes and with high trauma levels on their post-earthquake trauma level, coping skills, emotional eating situations and healthy lifestyle behaviors.

This research is a randomized controlled study that will be conducted in an online environment. The population of the research consists of students continuing their education in the Nursing Departments of Osmaniye Korkut Ata University, Fırat University Faculty of Health Sciences, and Ankara University Faculty of Nursing. The Post-Earthquake Trauma Level Determination Scale (PETLDS) will be administered to the entire population. The sample of the research will be stratified according to those who score high on the PETLDS (52 points and above) for each of the three universities and will be weighted according to the number of nursing students. Using a random sampling method, students will be assigned to experimental and control groups. It is planned to include a total of 80 students in the study, with 40 in the experimental group and 40 in the control group.

The study comprises five stages. The first stage, PREPARATION, involves obtaining ethical approval and permissions from universities, preparing data collection tools, and identifying scholarship recipients. The second stage is the development of the MOBILE AND WEB-BASED application. The third stage is the SITUATION ASSESSMENT stage. In this stage, the post-earthquake trauma level, coping skill level, emotional eating levels, and the status of healthy lifestyle behavior of students enrolled in the Nursing Departments of Fırat University, Osmaniye Korkut Ata University, and Ankara University will be determined using one of the quantitative data collection tools, PETLDS (Objectives 1, 2, 3, and 4). The fourth stage is the INTERVENTION stage, where the prepared training and applications will be implemented within the program (Objectives 5, 6, 7, and 8). The fifth stage is the EVALUATION stage, involving the collection of final test data and analysis.

In the proposed project, quantitative data will be collected through the Post-Earthquake Trauma Level Determination Scale, Earthquake Coping Strategies Scale, Healthy Lifestyle Behaviors Scale, and Emotional Eating Scale.

In this research project, psychosocial interventions will be implemented for students under the "Recovery Program" for a duration of 12 weeks. A mobile and web-based application program will be developed for the "Recovery Program", and all interventions will be conducted through this program. The Recovery Program will include activities such as screening of movies, laughter yoga, stress coping techniques training, progressive relaxation exercises, education on loss/grief processes, expressive art therapy applications, and training on healthy lifestyle behaviors. The proposed Project has a duration of 16 months and consists of 5 work packages.

It is anticipated that the proposed project will have significant social, economic, and scientific impacts. It is thought that the mobile and web-based application program to be implemented in this research will create a social support environment for students, provide professional psychosocial support, support the rehabilitation of students, set an example for post-traumatic intervention programs with different groups in the future, and can be included in national / provincial disaster action plans. The fact that the sample consists of students continuing their education in the same field will enhance interaction among students and contribute to their awareness of what can be done after a disaster in the future, thus also contributing to the identity of healthcare personnel. Among the suggested broader impacts of the proposed project are the publication of results in SSCI/SCI-E indexed journals and the training of researchers based on the findings of the research.

ELIGIBILITY:
Inclusion Criteria:

* Continuing education at all three universities where the research will be conducted
* The score obtained from the Post-Earthquake Trauma Level Determination Scale must be higher than the threshold value (52.38±5.05).

Exclusion Criteria:

• Students who have an existing psychiatric diagnosis and are in their final year will be excluded from the study.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-Earthquake Trauma Level Determination Scale (PETLDS) | At the end of week 1
  The scale developed by Tanhan and Kayri (2013) to quickly and easily evaluate PTSD symptoms in individuals, especially after the earthquake, consists of 20 items and 5 dimensions. These dimensions are Behavioral Problems, Excitatory Limitation, Affective, Cognitive Configuration and Sleep Problems. There are five-point Likert style expressions such as "I strongly disagree", "I slightly agree", "I moderately agree", "I strongly agree" and "I completely agree". Items 11 and 12 are reverse scored. The lowest score that can be obtained from the scale is 20 and the highest score is 100. Cronbach's alpha of the scale was found to be 0.87. Increasing scores from the scale indicate that individuals' level of exposure to earthquakes increases (Tanhan and Kayri, 2013).
Post-Earthquake Trauma Level Determination Scale (PETLDS) | At the end of week 12
  The scale developed by Tanhan and Kayri (2013) to quickly and easily evaluate PTSD symptoms in individuals, especially after the earthquake, consists of 20 items and 5 dimensions. These dimensions are Behavioral Problems, Excitatory Limitation, Affective, Cognitive Configuration and Sleep Problems. There are five-point Likert style expressions such as "I strongly disagree", "I slightly agree", "I moderately agree", "I strongly agree" and "I completely agree". Items 11 and 12 are reverse scored. The lowest score that can be obtained from the scale is 20 and the highest score is 100. Cronbach's alpha of the scale was found to be 0.87. Increasing scores from the scale indicate that individuals' level of exposure to earthquakes increases (Tanhan and Kayri, 2013).
Earthquake Stress Coping Strategies Scale (ESCSS) | At the end of week 1
  The scale, consisting of 16 items and 3 sub-dimensions, was developed by Yöndem and Eren (2008).
Earthquake Stress Coping Strategies Scale (ESCSS) | At the end of week 12
  The scale, consisting of 16 items and 3 sub-dimensions, was developed by Yöndem and Eren (2008).

SECONDARY OUTCOMES:
Health Lifestyle Behavior Scale | At the end of week 1
  Turkish validity Bahar et al. The scale made by has 52 items and six factors. These; spiritual development, interpersonal relationships, nutrition, physical activity, health responsibility and stress management. The overall score of the scale gives the score for healthy lifestyle behaviors. All items of the scale are positive. The rating is in the form of a 4-point Likert and is accepted as never (1), sometimes (2), often (3), and regularly (4). The lowest score for the entire scale is 52 and the highest score is 208. The Cronbach Alpha coefficient of the scale is 0.92; The reliability coefficients of the sub-dimensions are; Health responsibility was found to be 0.77, Physical Activity 0.79, Nutrition 0.68, Spiritual Development 0.79, Interpersonal Relations 0.80, Stress Management 0.64 (Bahar, 2008).
Health Lifestyle Behavior Scale | At the end of week 12
  Turkish validity Bahar et al. The scale made by has 52 items and six factors. These; spiritual development, interpersonal relationships, nutrition, physical activity, health responsibility and stress management. The overall score of the scale gives the score for healthy lifestyle behaviors. All items of the scale are positive. The rating is in the form of a 4-point Likert and is accepted as never (1), sometimes (2), often (3), and regularly (4). The lowest score for the entire scale is 52 and the highest score is 208. The Cronbach Alpha coefficient of the scale is 0.92; The reliability coefficients of the sub-dimensions are; Health responsibility was found to be 0.77, Physical Activity 0.79, Nutrition 0.68, Spiritual Development 0.79, Interpersonal Relations 0.80, Stress Management 0.64 (Bahar, 2008).
Emotional Eating Scale: | At the end of week 1
  The scale, validated in Turkish by Bilgen (2018), consists of four subscales and 30 items. The highest score from the scale can be 150 and the lowest score can be 30. Subdimensions of the scale; It consists of the dimensions of eating in situations of tension (11 items), eating to cope with negative emotions (10 items), self-control (6 items), and control in the face of stimuli (3 items). Cronbach's alpha number of the scale was found to be 0.95 (Bilgen, 2018)
Emotional Eating Scale: | At the end of week 12
  The scale, validated in Turkish by Bilgen (2018), consists of four subscales and 30 items. The highest score from the scale can be 150 and the lowest score can be 30. Subdimensions of the scale; It consists of the dimensions of eating in situations of tension (11 items), eating to cope with negative emotions (10 items), self-control (6 items), and control in the face of stimuli (3 items). Cronbach's alpha number of the scale was found to be 0.95 (Bilgen, 2018)

IPD SHARING:
Plan to Share IPD: No